CLINICAL TRIAL: NCT00186498
Title: Memantine as an Adjunctive Agent to Reduce Neurocognitive Deficits Following Unilateral ECT for the Treatment of a Severe Major Depressive Episode
Brief Title: Memantine to Reduce Neurocognitive Deficits Following Unilateral ECT for the Treatment of a Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Hugh Brent Solvason, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NAM-10
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Memantine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Oral Capsule (Placebo Comparator): Patients received a placebo capsule starting the day before ECT begins and while receiving ECT
  Interventions: Drug: Placebo Oral Capsule
- memantine (Experimental): Patients receive memantine starting the day before ECT begins and while receiving ECT
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: memantine — Patients received a memantine containing capsule starting the day before ECT begins and while receiving ECT
  Other Names: Nameda
  Arms: memantine
Drug: Placebo Oral Capsule — Patients received a placebo capsule starting the day before ECT begins and while receiving ECT
  Other Names: Sugar Pill
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this study is to determine whether taking the medication memantine reduces impairment of memory and attention associated with electroconvulsive therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the novel NMDA antagonist memantine, FDA approved for use in moderate to severe alzheimers dementia, may reduce the neurocognitive deficits associated with right unilateral ECT treatments in patients receiving ECT for a severe and relatively refractory Major Depressive episode.

Our hypothesis is that the use of an NMDA antagonist would reduce intracellular calcium levels, and glutamatergic stimulation during ECT. This reduction in excitatory stimulation during ECT would reduce hippocampal and prefrontal neuronal endangerment and dysfunction, thereby reducing cognitive impairment associated with right unilateral ECT treatments. We also hypothesize that ACTH and cortisol levels will correlate with neurocognitive impairment in placebo treated subjects, but not in the memantine treated individuals.

ELIGIBILITY:
Inclusion Criteria::

* Meets DSM-IV criteria for Major Depressive Disorder
* 18 to 75 years of age and able to provide legal consent
* Referred to Stanford ECT service by treating physician for unilateral electroconvulsive therapy with inpatient hospitalization
* Competed process for consenting to the clinical use of ECT according to California State law
* Females of childbearing potential will be required to use a double-barrier method of contraception, which includes foam and either condom and diaphragm, IUD, and/or implant during study.
 Exclusion Criteria:- Treatment with ECT in the 6 months prior to screening
* Meets criteria for drug or alcohol abuse or dependence in the 6 months prior to screening
* Use of alcohol or illegal drugs within seven days of randomization or during study. Patients may be excluded for use during a period greater than 7 days, per study physician's discretion
* Presence of unstable or untreated cardiovascular disease, hypertension, or endocrine disorder as determined by the investigator
* use of antipsychotic, antidepressant, or other prescription medications unless dose is stable for at least 7 days prior to randomization.
* Use of any investigational treatment within 30 days of randomization
* Previous allergic reaction to memantine or drugs of similar chemical structure.
* Women who are pregnant or breastfeeding are not advised to participate in the research study
* Any neurological disorder or organic brain condition that would confound neurocognitive testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-02; Primary Completion 2006-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Brent Solvason, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients over age 18 who are referred for ECT for unipolar or bipolar depression were screened and enrolled. All patients receive right unilateral lead placements, and otherwise the entire procedure would be delivered as per usual clinical care at our institution.
  Patients who sign an informed consent for this study were screened for eligibility.
Groups:
- Memantine: Patients receiving memantine for 2 days before ECT for a total of 30 days
- Placebo: Patients receiving placebo for 2 days before ECT for a total of 30 days
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 6 | 5
Completed | 4 | 3
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Memantine: Patients receive memantine starting the day before ECT begins and while receiving ECT
  memantine: Memantine vs placebo
- Placebo: Patients receive placebo starting the day before ECT begins and while receiving ECT
  memantine: Memantine vs placebo
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (13.1) | 42.5 (11.3) | 41.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Memantine Effect on CVLT Long Term Recall After Right Unilateral ECT Treatment.
Description: The California Verbal Learning Test Delayed Free Recall is a measure of episodic verbal learning and memory. These results are from the Free Recall subtest. In this test the subject must recall a list of 16 nouns after 20 minutes without cueing. It assesses auditory encoding, recall and recognition. Scores reflect the number of correct recall of the presented words, and scores are are then normalized by age. A higher score reflects better memory function.
Time Frame: 30 days
Population: The subjects enrolled in the study had signed a consent to receive ECT treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Memantine: Patients are randomized 1:1, memantine treatment is for 2 days before ECT for a total of 30 days
- Placebo: Patients are randomized 1:1, placebo treatment is for 2 days before ECT for a total of 30 days
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 10.17 (5.565) | 6.67 (4.590)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Test type: Superiority or Other; p = 0.006, Regression, Linear — Test of within subjects contrast: CVLT Long Delay Free Recall Time 1 (baseline) vs Time 2 (30 days): Placebo (F 4.093) p= 0.071; Memantine (F 35.042) p=0.006

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No